CLINICAL TRIAL: NCT02067845
Title: Pilot-testing a Group-level Intervention to Reduce Risk for Sexual Transmission of HIV/STIs Among Lesbian, Bisexual and Queer Women and Other Women Who Have Sex With Women in Calgary and Toronto
Brief Title: A Group-level Intervention to Reduce HIV/STI Risk for Women Who Have Sex With Women in Calgary and Toronto
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: The CIHR Social Research Centre in HIV Prevention (Unknown)
Responsible Party: Principal Investigator, Carmen Logie, MSW, PhD, Assistant Professor at the Factor-Inwentash Faculty of Social Work, University of Toronto, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CIHR SRC - 4487453
Record Dates: First submitted 2014-02-18; First posted 2014-02-20 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Safer Sex
Keywords: Lesbian, queer, bisexual women; HIV and STI prevention; Resilient coping; Sexual stigma; Depression; Safer-sex practices; Safer sex self-efficacy; HIV/STI knowledge and testing; Pilot-testing
MeSH Terms: conditions — Homosexuality, Female; Homosexuality; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pre-post test design (Other)
  Interventions: Behavioral: Adapted Many Men, Many Voices (3MV) group level intervention; Behavioral: A group-based HIV/STI prevention intervention for women who have sex with women

INTERVENTIONS:
Behavioral: Adapted Many Men, Many Voices (3MV) group level intervention — The intervention will adapt the Many Men, Many Voices (3MV) group level intervention for MSM to address individual and social determinants of HIV/STI risk and vulnerability. This intervention involves 6 consecutive 2-3 hours sessions conducted at a weekend retreat. We will have 1 retreat in Calgary and 1 retreat in Toronto; each retreat will include 20 persons.
  Based on the 3MV format, a draft template includes: Session 1: Intersectionality; Session 2: STI/HIV Prevention Among WSW and LBQ Women; Session 3: STI/HIV Risk Assessment and Prevention Options; Session 4: Relationship Issues; Session 5: Self-efficacy, Resilient Coping and Capacity for Change; Session 6: Social Support and Problem Solving to Maintain Change.
  Delivery methods include discussion, role-plays and risk-reduction planning.
Behavioral: A group-based HIV/STI prevention intervention for women who have sex with women

SUMMARY:
The limited research that exists suggests that lesbian, bisexual and queer (LBQ) women are at similar risk for sexually transmitted infections (STI) as heterosexual women. This is a particularly important area to address, as literature highlights the convergence of sexual stigma and gender-based sexual violence as elevating LBQ women's risk for HIV and STI infection. However, recent Statistics Canada data indicated that: lesbians reported significantly lower rates of Pap testing than heterosexual or bisexual women; lesbians and bisexual women had higher odds of not having a regular doctor than heterosexual women; and bisexual women had higher reported unmet health care needs than lesbian and heterosexual women. These differences highlight the importance of implementing and evaluating interventions to address STI risk among LBQ women; however, no published study exists of this nature. A STI prevention intervention will be implemented with groups of LBQ women and WSW in Toronto and Calgary. The study has 5 distinct components: 1) key informant interviews to inform the development of the intervention training manual and survey questionnaire, 2) pre-test; 3) intervention (6 group sessions during a weekend retreat); 4) post-test directly following intervention, and 5) follow-up post-tests at 6 and 12 weeks. The study hypothesis is that, compared to pre-intervention, participants who receive the group-based intervention will report an increase in sexually transmitted infections (STI) knowledge post-intervention. The secondary hypotheses are that, compared with pre-intervention, participants will demonstrate higher mean scores of (a) safer sex self-efficacy; (b) STI testing; (c) safer sex practices; (d) resilient coping, (e) self-esteem, (f) social provisions, (g) community connectedness and (h) access to health care. We anticipated that compared to pre-intervention, participants post-intervention would report lower mean scores of (a) depression and (b) internalized stigma.

DETAILED DESCRIPTION:
This is a single-centre pragmatic N-of-1 pilot study. The target population is LBQ women in Calgary and Toronto, Canada. The authors aim to recruit 40 participants using purposive peer-driven recruitment methods. LBQ women from agencies that serve LBQ women will deliver the intervention. A survey will be conducted at pre and post-intervention to evaluate the impact of the intervention. Paired-sample t-tests will be used to assess pre- and post- intervention differences in sexual risk behaviour outcomes (safer sex practices, safer sex self-efficacy), protective factors (resilient coping, HIV/STI knowledge and testing) and social-structural determinants (social support, access to health care, internalized sexual stigma) directly following the intervention and 3 months post-intervention. Logistic and linear generalized estimating equation (GEE) regression models will be used to assess intervention effects for the follow-up period of 3 months to control for repeated within-subject measurements.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified lesbian, bisexual, queer, or women who have sex with women
* Over 18 years old who
* Are capable of providing informed consent
* Are interested in attending a weekend retreat with 6 group sessions and 3 month follow up
* Live in the greater Calgary and Toronto area.

Exclusion Criteria:

* Below 18 years old
* Does not identify as lesbian, bisexual or queer or a WSW
* Insufficient interest/attention to attend the group sessions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
STI knowledge | 3 months
  Sexually Transmitted Disease Knowledge Questionnaire (STD-KQ)

SECONDARY OUTCOMES:
Safer sex self-efficacy | 3 months
  A modified Condom Use Self Efficacy Scale, for enhanced appropriateness for LBQ women
STI and HIV incidence | 3 months
  Self-reported HIV/STI testing history and incidence (lifetime and in past 3 months)
Safer sex practices | 3 months
  Safer Sexual Practices among Lesbian Women' Scale
Resilient coping | 3 months
  Brief Resilient Coping Scale
Social Provisions | 3 months
  Social Provisions Scale
Internalized sexual stigma | 3 months
  Revised Internalized Homophobia Scale (IHP-R)
Sexual stigma | 3 months
  Homophobia Scale
Depression | 3 months
  Patient Health Questionnaire 2
Access to care | 3 months
  Participants will responded to questions asking if they had ever received (i) an HIV test and (ii) an STI test (not including HIV). Participants also responded to questions asking if they had ever experienced the following barriers to accessing health care: (i) cost travel, (ii) cost medications and (iii) belief that their HCP was not comfortable with their sexual orientation. Follow up surveys will ask if participants had received an HIV or STI test in the past 4 weeks.
Self-Esteem | 3 months
  Rosenberg Self Esteem Scale

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Logie, PhD, Principal Investigator — University of Toronto, Factor-Inwentash Faculty of Social Work
Locations (2):
- Canada (2):
  - Faculty of Social Work, University of Calgary, Calgary, Alberta
  - University of Toronto, Factor-Inwentash Faculty of Social Work, Toronto, Ontario

REFERENCES:
- [Derived] Logie CH, Lacombe-Duncan A, Weaver J, Navia D, Este D. A Pilot Study of a Group-Based HIV and STI Prevention Intervention for Lesbian, Bisexual, Queer, and Other Women Who Have Sex with Women in Canada. AIDS Patient Care STDS. 2015 Jun;29(6):321-8. doi: 10.1089/apc.2014.0355. Epub 2015 Apr 13. PMID 25867642
- [Derived] Logie CH, Navia D, Rwigema MJ, Tharao W, Este D, Loutfy MR. A group-based HIV and sexually transmitted infections prevention intervention for lesbian, bisexual, queer and other women who have sex with women in Calgary and Toronto, Canada: study protocol for a non-randomised cohort pilot study. BMJ Open. 2014 Apr 23;4(4):e005190. doi: 10.1136/bmjopen-2014-005190. PMID 24760356